CLINICAL TRIAL: NCT05399199
Title: The Effect of Virtual Reality Distraction on Pain and Anxiety During Arteriovenous Fistula Puncture Among Hemodialysis Patients: Randomized Controlled Trial
Brief Title: Virtual Reality Distraction During Arteriovenous Fistula Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, mohamed elsayed hamed elzeky, lecturer, medical surgical nursing department, faculty of nursing, Mansoura university, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: mansU
Record Dates: First submitted 2022-05-22; First posted 2022-06-01 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-10

CONDITIONS: Pain Management; Hemodialysis; Virtual Reality
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Procedure: virtual reality distraction
- control group (No Intervention)

INTERVENTIONS:
Procedure: virtual reality distraction — study group patients will view VR scene for 6 minutes before puncture .It involves a soothing nature experience and calming background music. Patients in intervention group will not able to see the puncture procedure due to the VR glasses.
  Arms: study group

SUMMARY:
The cannulation of arteriovenous fistula is a painful procedure in hemodialysis patients. Previous studies have shown the effectiveness of virtual reality in reducing pain during needle-related procedures

DETAILED DESCRIPTION:
Patients undergoing hemodialysis experience anxiety and pain related to the insertion of hemodialysis needles, estimated 320 times in total per year. The pain experienced is mostly caused by needle insertion into a fistula. Pain control is one of the main nursing tasks. Pain relief leads to the acceptance of the procedure and ultimately enhances the patients' quality of life. The use of virtual reality to reduce pain and anxiety during the arteriovenous fistula cannulation procedure is based on the concept that the perception of pain can be controlled because an individual is able to process only a limited amount of information at once. As such, the use of virtual reality during painful procedures may serve as a distraction.

ELIGIBILITY:
Inclusion Criteria:

* patients who are under- going conventional hemodialysis three times a week
* hemodialysis period of one month or more
* having a healthy AVF access with good function
* welling to participate in study

Exclusion Criteria:

* patients who have psychiatric diseases
* panic disorder, anxiety disorder
* dysfunctional fistula
* vertigo, issues with sight, hearing, or perception
* or use painkillers within three hours before hemodialysis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Actual)
Dates: Start 2022-06-05 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
change in patients pain scores | will be measured at baseline and immediately after intervention (after 6 minutes of VR distraction)
  visual analogue scale which consists of a vertical line 100 mm long, one end of the line reads "No pain" and at the other is "Unbearable pain
change in patients anxiety scores | will be measured at baseline and immediately after intervention (after 6 minutes of VR distraction)
  STAI includes two subscales with 20 items each that assess state and trait anxiety .The State Anxiety Scale requires individuals to describe their feelings at a specific moment under specific circumstances, while the Trait Anxiety Scale requires them to describe the way they feel in general.

SECONDARY OUTCOMES:
change in patients satisfaction score | will be measured at baseline and immediately after intervention (after 6 minutes of VR distraction)
  . The patients will be asked to rate procedure satisfaction placing a mark on a 100-mm vertical visual analogue scale
change in patients heart rate | will be measured at baseline and immediately after intervention (after 6 minutes of VR distraction)
  checklist will be used to assess heart rate after puncture
change in patients respiratory rate | will be measured at baseline and immediately after intervention (after 6 minutes of VR distraction)
  checklist will be used to assess respiratory rate after puncture
change in patients systolic blood pressure | will be measured at baseline and immediately after intervention (after 6 minutes of VR distraction)
  checklist will be used to assess systolic blood pressure after puncture
change in patients diastolic blood pressure | will be measured at baseline and immediately after intervention (after 6 minutes of VR distraction)
  checklist will be used to assess diastolic blood pressure after puncture
change in patients Oxygen saturation (SpO2) | will be measured at baseline and immediately after intervention (after 6 minutes of VR distraction)
  checklist will be used to assess Oxygen saturation after puncture

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No